CLINICAL TRIAL: NCT02855099
Title: Can Rehabilitation After TAVI Precipitate Recovery and Improve Prognosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: could not find eligible patients
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Director. Research & development, Tel-Aviv Sourasky Medical Center, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TASMC-16-UC-0015-16-TLV-CTIL
Record Dates: First submitted 2016-07-24; First posted 2016-08-04 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CR group (Active Comparator): patients will be referred to our rehabilitation centre at the following week after the procedure, and assigned to a personalized rehabilitation program for duration of 3 month.
  Interventions: Other: Rehabilitation
- conservative group (No Intervention): No intervention

INTERVENTIONS:
Other: Rehabilitation — The duration on the rehabilitation will be 3 month and will be a multidisciplinary program that includes supervised physical activity
  Arms: CR group

SUMMARY:
Many patients we encounter a month post TAVI, still complain of having symptoms limiting their daily activity. The investigators set out to study whether rehabilitation strategy early after the procedure contributes to reduction of the physical disability these patients suffer from.

Cardiac rehabilitation (CR) is a well-established treatment in patients who underwent cardiac surgery. Patients after TAVI, are natural candidates for referral to exercise-based CR. Despite this, until 2013 no data have been available about the safety and the efficacy of a comprehensive rehabilitative period in these subjects. CR is a helpful tool to maintain independency for daily life activities and participation in socio-cultural life. despite these differences, both patient groups did benefit in the same way from a post-acute in-patient rehabilitation program as assessed by 6-Minute Walking Tests and FIM scores. Patients who were unable to walk and those were slow walkers at baseline experienced an improvement in functional status after TAVI, whereas the fast walkers did not improve and actually experienced a modest decrease in 6MWTD.It has been shown that patients referred for rehabilitation after TAVI are often very frail, with a high grade of functional impairment, dependence on others and high risk of clinical complications. During a rehabilitation program, based on a multidimensional assessment and intervention, most patients showed significant improvement in functional status, quality of life, and autonomy, which remained stable in the majority of subjects during mid-term follow-up.

To the investigators knowledge, no prospective study compared rehabilitation strategy to conservative treatment after TAVI. the investigators set off to test the investigators hypothesize that CR may help in the short and long term prognosis of these patients.

DETAILED DESCRIPTION:
Many patients we encounter a month post TAVI, still complain of having symptoms limiting their daily activity. The investigators set out to study whether rehabilitation strategy early after the procedure contributes to reduction of the physical disability these patients suffer from.

Cardiac rehabilitation (CR) is a well-established treatment in patients who underwent cardiac surgery. Patients after TAVI, are natural candidates for referral to exercise-based CR. Despite this, until 2013 no data have been available about the safety and the efficacy of a comprehensive rehabilitative period in these subjects. Nicola Russo et al. compared the safety and efficacy of a structured, exercise-based CR program in octogenarians after a traditional sAVR vs. TAVI, and concluded that a short-term, supervised, exercise-based CR is feasible, safe and effective in octogenarian patients after TAVI as well as after traditional surgery. An early CR program enhances independence, mobility and functional capacity and should be encouraged in all patients. Long-term effects and prognostic relevance should be evaluated in future studies. A similar comparison assessed the hypothesis that patients after TAVI benefit from CR, compared to patients after surgical aortic-valve replacement (sAVR). They too concluded that patients after TAVI benefit from cardiac rehabilitation despite their older age and comorbidities. CR is a helpful tool to maintain independency for daily life activities and participation in socio-cultural life. The same conclusion was made by Ivan Fauchère et al. letter to the editor - patients in the TAVI group were older and sicker than SAVR patients. Despite these differences, both patient groups did benefit in the same way from a post-acute in-patient rehabilitation program as assessed by 6-Minute Walking Tests and FIM scores.

Another study, drawn from a cohort of 484 patients with severe symptomatic AS who underwent TAVI, evaluated the association between physical performance as estimated by the 6-minute walk test distance (6MWTD) and long-term prognosis after TAVI. They found that compared with those with 6MWTD above the median value, those who were unable to walk experienced a higher rate of death after TAVI. In contrast, patients who were unable to walk and those were slow walkers at baseline experienced an improvement in functional status after TAVI, whereas the fast walkers did not improve and actually experienced a modest decrease in 6MWTD.

It has been shown that patients referred for rehabilitation after TAVI are often very frail, with a high grade of functional impairment, dependence on others and high risk of clinical complications. During a rehabilitation program, based on a multidimensional assessment and intervention, most patients showed significant improvement in functional status, quality of life, and autonomy, which remained stable in the majority of subjects during mid-term follow-up.

To the investigators knowledge, no prospective study compared rehabilitation strategy to conservative treatment after TAVI. the investigators set off to test our hypothesize that CR may help in the short and long term prognosis of these patients.

ELIGIBILITY:
Inclusion Criteria:

* All TAVI patients above the age of 75
* male or female
* undergoing the TAVI procedure between 1 March 2016 - 1 March 2017
* signed informed consent.

Exclusion Criteria:

* Unstable clinical condition - according to treating physician.
* Handicap before the procedure.
* Severe cognitive decline.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-07-23 (Actual); Study Completion 2017-07-24 (Actual)

PRIMARY OUTCOMES:
quality of life questionnaire | 3 months
6 min walk test | 3 months
  number of meters the patient walked for 6 minutes to test the physical performance by the patient.

IPD SHARING:
Plan to Share IPD: No